CLINICAL TRIAL: NCT01884961
Title: Radiotherapy As an Immunological Booster in Patients with Metastatic Melanoma or Renal Cell Carcinoma Treated with High-dose Interleukin-2: Evaluation of Biomarkers of Immunologic and Therapeutic Response
Brief Title: Radiotherapy As an Immunological Booster in Patients with Metastatic Melanoma or Renal Cell Carcinoma Treated with High-dose Interleukin-2
Acronym: IL2HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST172.03; 2012-001786-32 (EudraCT Number)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Renal Cell Cancer; Malignant Melanoma, Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm A (Experimental): Boost of radiotherapy + high dose IL-2 treatment: Three daily doses boost radiotherapy at 6-12 Gy to at least 1, and up to a maximum of 5, metastatic fields, will be administrated on days -4 -3 -2 or -3 -2 -1 before the first and the third cycle of IL-2 (Interleukin 2). The first day of administration of IL-2 of each cycle is the day +1.
  Treatment with IL-2 (dose 18 MIU/m2/day in 500cc by continuous IV (intravenous) infusion for 72 hours) will start on day +1 and will be administered every 3 weeks up to 4 cycles, than every 3-4 weeks for a further 2 cycles.
  Patients will be evaluated every 8 weeks with computed tomography to determine the response, and every 3 months after completion of treatment until death.
  Interventions: Other: Boost of radiotherapy + high dose IL-2 treatment

INTERVENTIONS:
Other: Boost of radiotherapy + high dose IL-2 treatment — Boost of radiotherapy + high dose IL-2 treatment

SUMMARY:
Title: Radiotherapy as an immunological booster in patients with metastatic melanoma or renal cell carcinoma treated with High-dose Interleukin-2: evaluation of biomarkers of immunologic and therapeutic response

Phase: Proof of Principle phase II study

Study Design: Single center, open-label trial to assess the immune response and potential biomarkers predictive of response

Study Duration:

Total duration: 36 months Enrollment: 20 months Treatment: 5 months per patient Follow-up every three months

Number of Subjects:

Mini-max two-stage Simon design:

• Step 1: 7 patients enrolled

If tumor antigen-specific immune response is observed in at least 3 patients:

• Step 2: recruitment of an additional 12 patients

DETAILED DESCRIPTION:
Title: Radiotherapy as an immunological booster in patients with metastatic melanoma or renal cell carcinoma treated with High-dose Interleukin-2: evaluation of biomarkers of immunologic and therapeutic response

Phase: Proof of Principle phase II study

Study Design: Single center, open-label trial to assess the immune response and potential biomarkers predictive of response

Study Duration:

Total duration: 36 months Enrollment: 20 months Treatment: 5 months per patient Follow-up every three months

Primary objectives:

1. to determine the tumor antigen-specific immune response induced by the treatment
2. to prospectively determine the predictive/prognostic value of pretreatment biological features in identifying patients who will benefit from HDIL-2-based therapy

Secondary end points:

1. Toxicity
2. Response Rate
3. Overall Survival.

Number of Subjects:

Mini-max two-stage Simon design:

• Step 1: 7 patients enrolled

If tumor antigen-specific immune response is observed in at least 3 patients:

• Step 2: recruitment of an additional 12 patients

Study Product, Dose, Route, Regimen and duration of administration:

Three daily doses boost radiotherapy (XRT) at 6-12 Gy to at least 1, and up to a maximum of 5, metastatic fields, will be administrated on days -4 -3 -2 or -3 -2 -1 before the first and the third cycle of IL-2. The first day of administration of IL-2 of each cycle is the day +1.

Treatment with IL-2 (dose 18 MIU/m2/day in 500cc by continuous IV infusion for 72 hours) will start on day +1 and will be administered every 3 weeks up to 4 cycles, than every 3-4 weeks for a further 2 cycles.

IL-2 will be withheld for refractory hypotension (hypotension where isotropic or vasoactive therapy is ineffective and that persists despite specific medical therapy set), anuria for > 24 hours, respiratory distress, confusion, sustained ventricular tachycardia, signs of myocardial ischemia or myocarditis, persistant metabolic acidosis, atrial fibrillation and documented systemic infection.

Patients will be evaluated every 8 weeks with computed tomography to determine the response, and every 3 months after completion of treatment until death (the time of disease progression and the initiation of alternative therapies will also be documented).

Statistical Methodology:

A minimax two-stage Simon design will be employed. A 40% immune response will preclude further study, whereas a 70% response rate will indicate that further study would be warranted. Using alfa and beta errors of 0.10, 7 patients will be enrolled during the first stage, and if an immune response is observed in at least 3 patients the study will go on, and an additional 12 patients will be treated. The treatments will be considered active if a tumor antigen-specific immune response is observed in 11 out of 19 patients treated. The analysis will be performed on an intention to treat population, i.e. all patients having received at least one cycle of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed non resectable stage III or IV advanced melanoma or Renal Cell Carcinoma (RCC).
2. Patients must have a minimum of two lesions and one of which must be measurable, (it can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan).
3. At least one tumor lesion accessible for bioptic sampling.
4. Prior lines (maximum 4) of chemotherapy, immunotherapy or biological therapy (e.g. inhibitors of B-Raf or c-Kit, Ipilimumab, etc.) for advanced disease are allowed (patients must have finished prior treatments at least 4 weeks before the first IL2 dose);
5. Male or Female, aged >= 18 years.
6. Life expectancy of greater than 3 months.
7. ECOG performance status <=1
8. Patients must have normal organ and marrow function as defined below:

   * leukocytes >=3,500/microL
   * absolute neutrophil count >=1,500/microL
   * platelets >= 100,000/microL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal
   * creatinine < 1,2 mg/dl
   * haemoglobin > 9.0 gm/dl
   * ECG and echocardiogram within normal institutional limits
   * Pulmonary function tests within normal institutional limits (to be performed only in patients with lung metastases or history of impaired lung function)
9. no contraindication for the use of vasopressor agents
10. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
11. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Patient with stage I or II melanoma or RCC
2. Patients who have had chemotherapy or radiotherapy or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2 or other agents used in the study.
6. Any autoimmune disease which could be exacerbated by IL-2
7. A medical illness requiring chronic treatments with corticosteroids or other immunosuppressive agents
8. A history of significant cardiovascular disease, including myocardial infarction, congestive heart failure, primary cardiac arrhythmias, angina pectoris or cerebrovascular accident
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);
11. HIV-positivity, whether or not symptomatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
immunological efficacy | 3 years
  Determination of the immunological efficacy of the combined RT (radiotherapy)/HDIL-2 (high dose Interleukin 2) treatment in terms of ability of the treatment to enhance the proportion of circulating immune effectors specific for tumor antigens known to be expressed in RCC (Renal Cell Carcinoma) and/or melanoma
Biomarkers predictive value for treatment benefit | 3 years
  Determination of the predictive value of pretreatment biomarkers in identifying patients who will benefit from combined RT/HDIL-2 treatment

SECONDARY OUTCOMES:
Toxicity from the time of their first treatment with HD 2. | 3 years
  Evaluation of safety and tollerability of the experimental treatment. The percentage of patients reporting an Adverse Event (AE) up to 30 days after HD-IL-2 treatment will be tabulated with 95% confidence intervals, by type of AE. The overall rate of grade 3-4 related AE will be computed.
Response Rate | 3 years
  Evaluation of the response rate of treated patients
Overall Survival | 3 years
  Evaluation of the overall survival of treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ridolfi, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (1):
- UO Oncologia Medica, IRCCS IRST, Meldola (FC), FC, Italy

REFERENCES:
- [Derived] Ridolfi L, de Rosa F, Ridolfi R, Gentili G, Valmorri L, Scarpi E, Parisi E, Romeo A, Guidoboni M. Radiotherapy as an immunological booster in patients with metastatic melanoma or renal cell carcinoma treated with high-dose Interleukin-2: evaluation of biomarkers of immunologic and therapeutic response. J Transl Med. 2014 Sep 23;12:262. doi: 10.1186/s12967-014-0262-6. PMID 25245327